CLINICAL TRIAL: NCT00537836
Title: A Double-blind, Randomized, Placebo and Active Controlled, Multicenter Study to Investigate Efficacy and Safety After Oral Administration of 2 and 3 mg ZK 283197, 1 mg 17ß-estradiol and Placebo Once Daily for 8 Weeks in Postmenopausal Women With Hot Flushes
Brief Title: ZK283197 for Treatment of Vasomotor Symptoms
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91544; 2007-001791-36 (EudraCT Number); 310781 (Other: Company internal)
Record Dates: First submitted 2007-09-28; First posted 2007-10-01 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Vasomotor System
Keywords: Hot flushes; Therapy of hot flushes; 17ß-estradiol (E2); Hormone replacement therapy
MeSH Terms: conditions — Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- ZK 283197, 3 mg (Experimental): Postmenopausal women with hot flushes received 3 mg (3 x 1 mg tablets) ZK 283197, administered orally once daily over 8 weeks
  Interventions: Drug: BAY 86-5310 (ZK 283197)
- Matching placebo (Placebo Comparator): Postmenopausal women with hot flushes received placebo (3 tablets) orally once daily over 8 weeks
  Interventions: Drug: Placebo
- ZK 283197, 2 mg (Experimental): Postmenopausal women with hot flushes received 2 mg (2 x 1 mg tablet) ZK 283197 plus 1 placebo tablet, once daily orally over 8 weeks
  Interventions: Drug: BAY 86-5310 (ZK 283197)
- 17ß-estradiol (Active Comparator): Postmenopausal women with hot flushes received 1 mg (2 x 0.5 mg tablet) 17ß-estradiol plus 1 placebo tablet, once daily orally over 8 weeks
  Interventions: Drug: 17ß-estradiol

INTERVENTIONS:
Drug: BAY 86-5310 (ZK 283197) — 3 mg (3 x 1 mg tablet) or 2 mg (2 x 1 mg tablet) ZK 283197 in respective treatment group, once daily p.o. over 8 weeks
  Arms: ZK 283197, 2 mg; ZK 283197, 3 mg
Drug: Placebo — Placebo, once daily p.o. over 8 weeks
  Arms: Matching placebo
Drug: 17ß-estradiol — 1 mg (2 x 0.5 mg tablet) 17ß-estradiol, once daily p.o. over 8 weeks
  Arms: 17ß-estradiol

SUMMARY:
The primary goal of the planned study is to investigate the efficacy and safety of ZK 283197 in the dosage of 2 and 3 mg ingested once daily during a period of 8 weeks for the treatment of hot flushes. In order to be able to assess the efficacy of the test substance, this is compared with the efficacy of 1 mg Estradiol and placebo. The comparator Estradiol is a certified hormone preparation, which is already used for the treatment of hot flushes as standard treatment. After passing the screening, volunteers will start with a run-in phase followed by a 8 weeks treatment and a follow-up phase. 112 postmenopausal women with hot flushes and without relevant prior diseases will participate in three European countries (2 study sites in Germany, 1 study site in Great Britain and 1 study site in The Netherlands) in this study.

ELIGIBILITY:
Inclusion Criteria:

* Women with at least 35 moderate to severe hot flushes in seven consecutive days
* Body mass index (BMI) : 20 - 30 kg/m² (inclusive)
* Postmenopausal status

Exclusion Criteria:

* Contraindication for use for hormonal therapy
* Prior hysterectomy
* Hormonal therapy or intrauterine hormone releasing device within 4 weeks prior to study entry or any long-acting injectable or implant up to 6 months prior to study entry
* Repeated intake of medications affecting study aim

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2007-10; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Relative change in frequency of moderate to severe hot flushes per week between baseline and Week 8 of the treatment phase | Between baseline and Week 8 of the treatment phase

SECONDARY OUTCOMES:
Number of participants with adverse events | From Week 1 of treatment until end of Follow-up period (approximately 12 weeks)
Exposure-response relationship | At week 8
  A generalized linear model was applied to explore the dependence of the number of hot flushes in Week 8 to (i) the dose of ZK 283197, (ii) the AUC of ZK 283197, (iii) the maximum concentration Cmax of ZK 283197 and (iv) the average concentration Cave of ZK 283197
Change from baseline to all treatment weeks in frequency and severity of moderate to severe hot flushes | From baseline up to 8 weeks
Change from baseline to all treatment weeks in severity and frequency of all hot flushes | From baseline up to 8 weeks
Trough levels at every visit | Before 1st administration and at Week 1, 2, 4, 6 and 8
AUC(0-24h) | Pre-dose and up to 24 h post-dose (measured between Week 4-8)
  Area under the curve from administration to 24 h after administration
Cmax | Pre-dose and up to 24 h post-dose (measured between Week 4-8)
  Maximum serum concentration
tmax | Pre-dose and up to 24 h post-dose (measured between Week 4-8)
  Time to reach maximum drug concentration
Cmin | Pre-dose and up to 24 h post-dose (measured between Week 4-8)
  Minimum serum concentration
Cave | Pre-dose and up to 24 h post-dose (measured between Week 4-8)
  Average serum concentration
Vaginal cytology | Between baseline and Week 8
  The epithelial maturation index/value and the karyopycnotic index were assessed
Endometrial thickness | Fom baseline to Week 8
  Transvaginal ultrasound was performed to demonstrate the absence of relevant endometrium growth
Endometrial histology | Between baseline and Week 8

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (3):
- Berlin, State of Berlin, Germany
- Groningen, Netherlands
- Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/